CLINICAL TRIAL: NCT04052880
Title: A Phase 2 Study of Subcutaneous Daratumumab in Combination With Dose-Attenuated Bortezomib, Lenalidomide, and Dexamethasone in Elderly Newly Diagnosed Multiple Myeloma Patients
Brief Title: Study of SubQ Dara With Dose-Attenuated Bortezomib, Lenalidomide, Dexamethasone in Elderly NDMM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Larysa Sanchez (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor-Investigator, Larysa Sanchez, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 19-0944
Record Dates: First submitted 2019-08-02; First posted 2019-08-12 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Newly Diagnosed Multiple Myeloma
Keywords: Multiple myeloma; Newly diagnosed multiple myeloma; Myeloma; Elderly; Daratumumab
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — daratumumab; Bortezomib; Lenalidomide; Dexamethasone; ixazomib

STUDY DESIGN:
Intervention Model Description: All subjects will receive initial therapy with 12 cycles of daratumumab in combination with dose-attenuated bortezomib, lenalidomide and dexamethasone (VRd). Maintenance treatment cycles are 28 days in duration with daratumumab and either lenalidomide or ixazomib. The choice of maintenance therapy will be based on cytogenetic risk status at diagnosis. For patients with high-risk MM defined by FISH with t(4;14) only; maintenance therapy will consist of daratumumab with ixazomib. For all other patients, maintenance therapy will consist of daratumumab with lenalidomide. All subjects will continue maintenance treatment until disease progression, except maintenance daratumumab will be discontinued after 2 years if subjects remain on maintenance treatment at that time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Daratumumab with dose-attenuated VRd (Experimental): SubQ Daratumumab with Dose-Attenuated VRd
  Interventions: Drug: Daratumumab; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone; Drug: Ixazomib

INTERVENTIONS:
Drug: Daratumumab — Daratumumab 1800 mg will be delivered by subcutaneous injection given through a syringe and needle by a manual push over approximately 3 to 5 minutes. Doses will be administered at alternating locations on the abdomen. Daratumumab will be administered weekly during treatment in Cycles 1 to 2, every 2 weeks during cycles 3-6, and every 4 weeks thereafter.
Drug: Bortezomib — Subjects will receive 1.3 mg/m2 bortezomib as a subcutaneous infusion on Days 1, 8, and 15 during the 28-day cycles.
Drug: Lenalidomide — In Cycles 1 through 12, lenalidomide will be self-administered at a dose of 15 mg orally each day on Days 1 through 21 of each 28-day cycle.
  For subjects with CrCl 30-60mL/min, lenalidomide will be reduced to 10mg daily, and for subjects with CrCl 15-30 mL/min, lenalidomide will be reduced to 5mg daily.
  In maintenance phase: lenalidomide will be administered at one dose level below Cycles 1-12 dosing ie 10 mg orally daily.
  In maintenance, for subjects with CrCl 30-60 mL/min, lenalidomide will be reduced to 5 mg daily during maintenance treatment, and for subjects with CrCl 15-30 mL/min, lenalidomide will be reduced to 5 mg every other day during maintenance treatment.
Drug: Dexamethasone — Dexamethasone will be self-administered orally at a total dose of 20 mg weekly during cycles.
  However, the dexamethasone 20 mg oral or IV (only if oral is not available) dose administered as a preinfusion medication on daratumumab infusion days replaces the oral dexamethasone dose for that day. Dexamethasone will be administered until the subject experiences disease progression or unacceptable toxicity.
  In the maintenance phase, dexamethasone/steroid premedications may be tapered or discontinued in the absence of daratumumab related infusion reactions/based on patient tolerance. In the event of persistent daratumumab related infusion reactions, the least amount of steroid premedications needed to prevent the same may be used.
Drug: Ixazomib — During maintenance treatment, if choice of maintenance therapy includes ixazomib, ixazomib will be administered at 3 mg orally daily on Days 1,8, and 15 of each cycle. For subjects with CrCl 15-30 mL/min, ixazomib will be reduced to 2.3 mg once per week during maintenance treatment.

SUMMARY:
This is a single center, open-label, phase 2 study in elderly (age ≥ 70) subjects with newly diagnosed multiple myeloma who are transplant ineligible. Subjects will receive subcutaneous daratumumab, dose-attenuated bortezomib, revlimid, and dexamethasone until confirmed disease progression, discontinuation of study treatment due to unacceptable drug toxicity, or other reasons. Throughout the study, subjects will be monitored closely for adverse events, laboratory abnormalities, and clinical response.

DETAILED DESCRIPTION:
This is a single center, open-label, phase 2 study in elderly (age ≥ 70) subjects with newly diagnosed multiple myeloma who are transplant ineligible. The main study consists of the following phases: a 28-day screening phase; followed by initial therapy with 12 cycles of daratumumab in combination with dose-attenuated VRd; and a maintenance phase that starts after Cycle 12 of therapy. Cycles are 28 days in length. Treatment can continue until disease progression or unacceptable toxicity. After 12 cycles of initial therapy, maintenance therapy will begin with 28 day cycles of daratumumab with either lenalidomide or ixazomib and the choice of maintenance therapy will be based on cytogenetic risk status at diagnosis. All subjects will continue maintenance treatment until disease progression, except maintenance daratumumab will be discontinued after 2 years if subjects remain on maintenance treatment at that time. All subjects will be followed in the longterm follow-up for at least 1 year after last dose of study treatment and will continue until death, withdrawal of consent for study participation, or the end of study definition is met. The end of study is defined as when all subjects have completed at least 1 year of long-term follow up and until death, withdrawal of consent for study participation, or 5 years after first patient begins daratumumab therapy, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, untreated, symptomatic MM as defined by standard criteria. Clonal bone marrow plasma cells >10% or biopsy-proven bony or extramedullary plasmacytoma* and any one or more of the following myeloma-defining events:

  * Evidence of end-organ damage that can be attributed to the underlying plasma cell proliferative disorder, specifically:

    * Hypercalcemia: serum calcium >0.25 mmol/L (> 1mg/dL) higher than the upper limit of normal or > 2.75 mmol/L (>11 mg/dL) and/or,
    * Renal insufficiency: creatinine clearance <40 mL per min or serum creatinine >177 µmol/L (>2 mg/dL) and/or,
    * Anemia: hemoglobin value of >20 g/L (>2g/100 mL)below the lower limit of normal, or a hemoglobin value <100 g/L (10g/100 mL) and/or,
    * Bone lesions: one or more osteolytic lesions on skeletal radiography, CT, or PET-CT (if bone marrow has less than 10% clonal plasma cells, more than one bone lesion is required to distinguish from solitary plasmacytoma with minimal marrow involvement)
    * Any one or more of the following biomarkers of malignancy:

      * Clonal bone marrow plasma cell percentage** (clonality should be established by showing kappa/lambda-light-chain restriction on flow cytometry, immunohistochemistry, or immunofluorescence. Bone marrow plasma cell percentage should preferably be estimated from a core biopsy specimen; in case of a disparity between the aspirate and core biopsy, the highest value should be used ≥60% or
      * Serum free light chain (FLC) ratio greater than or equal to 100 provided involved FLC level is 100 mg/L or higher, or
      * More than one focal lesion on MRI*** (Each focal lesion must be 5 mm or more in size.
* Age ≥ 70 and ineligible for autologous hematopoietic stem cell transplantation (defined as age, ≥ 80 or age < 80 with cardiac/pulmonary/ or other comorbidities deemed by investigator likely to have a negative impact on tolerability of high dose chemotherapy with stem cell transplantation).
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Patients must have measurable disease defined by at least 1 of the following 3 measurements:

  * Serum M-protein > 1 g/dL (10 g/L) or > 0.5 g/dL if IgA
  * Urine M-protein > 200 mg/24 hours.
  * Serum free light chain assay: involved free light chain level >10 mg/dL (> 100 mg/L) provided the serum free light chain ratio is abnormal
* Due to the teratogenicity of lenalidomide and the lack of adequate reproductive toxicity data for daratumumab, if a male subject is sexually active with a woman of child bearing potential, in addition to the user independent highly effective method of contraception, a male or female condom with or without spermicide, diaphragm, or cervical cap is required. Male condom and female condom should not be used together (due to risk of failure with friction).
* During the study (including during dose interruptions), and for 4 weeks following discontinuation of lenalidomide, and if receiving daratumumab, for 3 months after the last dose, in addition to the user independent highly effective method of contraception (even if he has undergone a successful vasectomy), a man:

  1. Who is sexually active with a woman of childbearing potential must agree to use a barrier method of contraception (ie, latex or synthetic condom with spermicidal foam/gel/film/cream/suppository)
  2. Who is sexually active with a woman who is pregnant must use a latex or synthetic condom.
  3. Must agree not to donate sperm
* Willing and able to adhere to the prohibitions and restrictions specified in this protocol and referenced in the informed consent form (ICF)
* Must sign an ICF (or their legally acceptable representative must sign) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study.

Exclusion Criteria:

* Peripheral neuropathy > Grade 2 or >Grade 1 with pain on clinical examination during the Screening period.
* Kidney failure with CrCl ≤ 15 mL/min by Cockfraft Gault
* Significant cardiac disease as determined by the investigator including:

  1. Known or suspected cardiac amyloidosis
  2. Congestive heart failure of Class III or IV of the NYHA classification
  3. Uncontrolled angina, hypertension or arrhythmia
  4. Myocardial infarction in the past 6 months
  5. Any uncontrolled or severe cardiovascular disease
  6. QTc > 470 milliseconds (msec) on a 12-lead ECG obtained during the Screening period. If a machine reading is above this value, the ECG should be reviewed by a qualified reader and confirmed on a subsequent ECG or by manual calculation.
* Prior cerebrovascular event with persistent neurologic deficit.
* Subject is:

  1. Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using realtime polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
  2. Seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy).
* Human immunodeficiency virus infection
* Any medical conditions that, in the investigator's opinion, would impose excessive risk to the subject.
* Prior or concurrent malignancy, except for the following:

  1. Adequately treated basal cell or squamous cell skin cancer
  2. Cervical carcinoma in situ
  3. Adequately treated Stage I or II cancer from which the subject is currently in complete remission.
  4. Or any other cancer from which the subject has been disease-free for ≥ 3 years
* Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of study drug, including difficulty swallowing.
* Males sexually active with females of childbearing potential who do not agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form (ICF) through 90 days after the last dose of study drug, or do not agree to practice true abstinence.
* Central nervous system involvement.
* Diagnosis of primary amyloidosis (with the exception of patients whose amyloidosis has been documented as a complication of MM, who will be evaluated on a case-by-case basis for trial participation).
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study drug administration.
* Known chronic obstructive pulmonary disease with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal (for subjects > 65 years old FEV1 <50% or DLCO <50%). Note: FEV1 testing is required for subjects suspected of having chronic obstructive pulmonary disease and subjects must be excluded if FEV1 <50% of predicted normal.
* Known moderate or severe persistent asthma within the past 2 years or currently has uncontrolled asthma of any classification. Note: Subjects who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed in the study.
* Persistent corrected serum calcium ≥ 14 mg/dL within 2 weeks of enrollment (despite appropriate measure such a short course of steroids, bisphosphonates, hydration, calcitonin).
* Absolute neutrophil count < 1000 cells/mm3. No growth factors allowed within 1 week of enrollment.
* Platelets < 75,000 cell/mm3 (75 x 109/L). Qualifying laboratory value must occur at most recent measurement before enrollment and must be no more than 14 days before enrollment. No transfusions are allowed within 72 hours prior to study drug administration.
* Hemoglobin < 8 g/dL. Qualifying laboratory value must occur at most recent measurement before enrollment and must be no more than 14 days before enrollment. No transfusions are allowed within 72 hours before qualifying laboratory value.
* Total bilirubin > 1.5 x ULN, unless known have Gilbert's syndrome in which case 3 x ULN).
* AST or ALT ≥ 3 x ULN.
* Major surgery or radiation therapy within 14 days before study drug administration.
* Kyphoplasty or vertebroplasty within 1 week of enrollment.
* Administration of Anti-myeloma chemotherapy, biological, immunotherapy, or investigational agent (therapeutic or diagnostic) within 3 weeks before enrollment; however, a cumulative dose of ≤ 160 mg dexamethasone or equivalent during screening is permitted.
* NSAIDs, IV contrast, aminoglycosides, or other potentially nephrotoxic drugs within 2 weeks of enrollment, except aspirin.
* Known hypersensitivity to bortezomib, lenalidomide, dexamethasone, or daratumumab

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2019-10-24 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Responses: VGPR or better | At the end of cycle 8, each cycle is 28 days
  ≥ VGPR rate after 8 cycles of therapy, defined as the proportion of subjects who have achieved VGPR or better, according to the IMWG criteria.

SECONDARY OUTCOMES:
Overall Response Rates | Within a year
  ORR (≥PR), CBR (≥SD), ≥CR, and sCR rates defined as the proportion of subjects who achieve each of these response categories (or better response category) according to the IMWG criteria
Duration of ORR (≥PR), ≥VGPR, ≥CR, and sCR | Within two years
  Defined as the duration from the date of initial attainment of a response category (or better response category), according to the IMWG criteria, to the date of first documented evidence of relapse from CR (or sCR) or progressive disease (PD)
Time to Overall Response Rate | Within a year
  Defined as the duration from the date of initial therapy to the date of attainment of a response category and was subsequently confirmed by a repeated measurement as required by the IMWG criteria
Time to Progression | Within 2 years
  Defined as the duration from the date of initial therapy to the date of first documented evidence of progressive disease according to the IMWG criteria
Progression Free Survival | Within 5 years
  Defined as the duration from the date of initial therapy to the date of first documented evidence of PD or death, whichever comes first
Overall Survival | Within 5 years
  Defined as the duration from the date of initial therapy to the date of the subject's death.
Number of Adverse Events | Within 5 years
  To assess safety and tolerability using the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE Version 4.03)

CONTACTS AND LOCATIONS:
Overall Officials: Larysa Sanchez, Principal Investigator — Icahn School of Medicine at Mount Sinai; Sundar Jagannath, MBBS, Study Director — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No